CLINICAL TRIAL: NCT03922698
Title: Potential Impact of Neuroimmune and Autophagic Alterations on the Progression and Severity of Human Atherosclerotic Process
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Giuseppe Lembo, Full Professor, MD, PhD, Neuromed IRCCS
Other Study IDs: LMB06
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Carotid Atherosclerosis
Keywords: atherosclerotic plaque; autonomic nervous system; immune system; autophagy
MeSH Terms: conditions — Carotid Artery Diseases; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and serum, bioptic tissue (atherosclerotic plaque)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case Group: Patients who undergo surgical intervention of carotid trombo-endo-arterectomy at the Department of Vascular Surgery of the IRCCS Neuromed, with specific inclusion/exclusion criteria
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions - observational study

SUMMARY:
The hypothesis of this study is that neural regulations of the atherosclerotic plaque, identified in the murine model of atherosclerosis, could also exist in human pathology. The dysregulation status of the autonomic nervous system is typical of several cardiovascular diseases, but the role it exerts in the modulation of important mechanisms at the basis of the atherosclerotic process progression has not been investigated yet. The main aim of this study will be to investigate, in the atherosclerotic plaque, the alterations of inflammatory and immune processes, the neural modulations and the presence of dysregulations of the autophagic process. The investigators will also associate the potential presence of neural modulations of the plaque to its stability/instability, from a clinical-translational point of view. Finally, the investigators aim at providing a solid basis for the development of novel therapeutic strategies, which could reduce the elevated health and welfare costs for the clinical management of cardiovascular pathologies such as atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 45 and ≤ 90 years;
* patients with severe (70-99%) carotid stenosis, diagnosed with color doppler echography or angio-MRI or angiography;
* written informed consent.

Exclusion Criteria:

* carotid stenosis <70% at carotid bifurcation or diagnosed with color doppler echography or angio-MRI or angiography;
* severe neoplasia;
* participation to other clinical trial, ongoing or terminated less than one month before enrolment in this study.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from patients who will undergo to surgical intervention of carotid trombo-endo-arterectomy at the Department of Vascular Surgery of the IRCCS Neuromed, accordingly to the following inclusion/exclusion criteria. Approximately 50 subjects of both genders will be included in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of the neuro-modulation of immune system in atherosclerosis | At enrollment
  Immunohistochemistry and immunofluorescence of the autonomic nervous and immune systems in the atherosclerotic plaque, and flow cytometry analysis of circulating immune cells.
Characterization of the autophagic process and correlation with neural modulations of the stability/instability plaque | At enrollment
  Expression of autophagic markers and immunohistochemical analysis of the atherosclerotic plaque.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Lembo, MD, PhD, Principal Investigator — IRCCS Neuromed; Giacomo Frati, MD, PhD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: No